CLINICAL TRIAL: NCT07096453
Title: CMVIG Prophylaxis in Belatacept Conversion Kidney Transplant Recipients: a PK Pilot Study
Brief Title: CMVIG Prophylaxis in Belatacept Conversion Kidney Transplant Recipients
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SURG-2024-32817
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Kidney Transplant; Complications; CMV
Keywords: Kidney transplant; CMV prevention
MeSH Terms: interventions — cytomegalovirus-specific hyperimmune globulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Single Dose, Day 0 (Experimental): CMVIG 150 mg/kg x 1 at Day 0. Belatacept will be administered per standard of care (IV infusion over 30 minutes in an outpatient specialty infusion center). Cytogam will be administered according to the assigned dosing regimen starting 30 minutes after completion of Belatacept infusion.
  Interventions: Drug: Cytogam
- Two Doses, One Week (Experimental): CMVIG 150 mg/kg x 2. Dose #1: Day 0, Dose #2: Day 7. Belatacept will be administered per standard of care (IV infusion over 30 minutes in an outpatient specialty infusion center). Cytogam will be administered according to the assigned dosing regimen starting 30 minutes after completion of Belatacept infusion.
  Interventions: Drug: Cytogam
- Two Doses, Four Weeks (Experimental): CMVIG 150 mg/kg x 2. Dose #1: Day 0, Dose #2: Day 28. Belatacept will be administered per standard of care (IV infusion over 30 minutes in an outpatient specialty infusion center). Cytogam will be administered according to the assigned dosing regimen starting 30 minutes after completion of Belatacept infusion.
  Interventions: Drug: Cytogam

INTERVENTIONS:
Drug: Cytogam — Cytogam is used for the prevention of cytomegalovirus (CMV) disease in kidney, lung, liver, pancreas, heart and bone marrow transplantation. We do not yet have data about how much cytogam reduces CMV in blood, or how quickly it reduces CMV in blood.

SUMMARY:
The purpose of this study is to study how CMVIG interacts with the body and to see if it might work to prevent kidney transplant patients from becoming infected with CMV.

ELIGIBILITY:
Inclusion Criteria:

* Adult (18-70 year old) kidney transplant recipients
* Patients transitioning from conventional CNI-based immunosuppression to co-stimulatory blockade (belatacept) immunosuppression OR patients who are stable on belatacept immunosuppression at the time of initial CYTOGAM infusion
* CMV Ig Seronegative Recipient who received a CMV Ig seropositive Donor
* EBV IgG Positive

Exclusion Criteria:

* Pregnant people
* Subjects unwilling to sign consent and complete follow up visits
* Subjects with IgA immunodeficiency
* Subjects who are receiving IgG therapy or who have received IgG therapy within two months of study enrollment
* Patients who do not speak English and would need a translator and translated consent materials in order to obtain informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Anti-CMV IgG antibody level: Day 0 | Day 0, pre-infusion
  Measured with ELISA testing
Anti-CMV IgG antibody level: Day 7 | Day 7
  Measured with ELISA testing
Anti-CMV IgG antibody level: Day 14 | Day 14
  Measured with ELISA testing
Anti-CMV IgG antibody level: Day 21 | Day 21
  Measured with ELISA testing
Anti-CMV IgG antibody level: Day 28 | Day 28
  Measured with ELISA testing
Anti-CMV IgG antibody level: Day 56 | Day 56 after last dose of CMVIG
  Measured with ELISA testing

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Humphreville, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No